CLINICAL TRIAL: NCT00224341
Title: Arrhythmia Restart Prevention and RatE STabilization in Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitatron France (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ARREST-AF
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-09

CONDITIONS: Sick Sinus Syndrome; Brady-Tachy Syndrome
Keywords: Pacemaker; Atrial Fibrillation; Prevention pacing; Algorithms; Sick sinus syndrome + Atrial Fibrillation
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

INTERVENTIONS:
Device: Pacemaker Vitatron Selection 9000
Device: Pacemaker Vitatron T70

SUMMARY:
The objective of this trial is to show the therapeutic efficacy of the preventive pacing therapies of the Selection 9000 and Vitatron T70 DR pacemakers, dedicated to handle atrial fibrillation (AF). Two new algorithms (post-AF response and ventricular rate stabilization [VRS]) will be assessed in a combined pathway, compared to a control group. The efficacy of the overall available therapies to prevent AF and its symptoms will then be assessed also.

DETAILED DESCRIPTION:
Due to anti-arrhythmic pharmacological drugs failure to suppress atrial fibrillation (AF), interest towards preventive pacing treatments is increasing. The importance of this option in the panoply of the preventive tools is fully justified, only by considering the insufficiency, the complexity, or the poor reproducibility of the other non-pharmaceutical approaches.

Preventive pacing therapies rely on their potential effect on different onset modalities emphasized by previous studies, and more generally by stabilizing atrial tissue when potential triggers are appearing.

On top of that, cardiac stimulator can deliver these therapies when identifying these triggers but also can offer incomparable diagnostic tools, in terms of sensitivity, specificity and continuity in the monitoring.

Four preventive pacing therapies have already been evaluated, the objective of this study is to show the clinical benefit brought by the new features of the Selection 9000 / Vitatron T70 DR.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented atrial fibrillation: at least one episode of paroxysmal AF documented 6 months prior to inclusion, lasting more than one minute
* Patient with a brady-tachy syndrome or a sick sinus syndrome, with a permanent pacing indication
* Atrial lead with a tip-to-ring interval equal to or less than 12 mm
* Patient who agrees with and has signed the informed consent

Exclusion Criteria:

* Permanent AF
* AF related to a reversible cause
* One electrical cardioversion 6 months prior to inclusion
* Unstable angina
* Myocardial infarction (MI) less than 3 months
* Planned cardiac surgery or performed in the last 3 months
* Congestive heart failure, New York Heart Association (NYHA) class IV
* Life expectancy less than 18 months
* Patient participating in other studies
* Patient not able to follow the FU calendar
* Less than 18 years of age
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-11; Study Completion 2006-11

PRIMARY OUTCOMES:
Show clinical benefit of post-AF response and VRS algorithms, when combined versus compared with a control group: In a conventional dual chamber (DDD) configuration
In a configuration including all the preventive pacing therapies of the device
The primary endpoint is the atrial fibrillation burden.

SECONDARY OUTCOMES:
Assess the effect of post-AF response and VRS, when combined versus compared with a control group, in a conventional DDD configuration and another configuration which includes all PPT, on: Number (Nb) of hospitalizations
Nb of cardioversions
Symptom score
Restarts
Daily incidence of AF
Mean sinus rhythm duration
Assess clinical benefit of the overall AF therapies, as compared with the first four algorithms of the previous device (one continuous overdrive +3 triggered overdrive), on the same outcomes as above and AF burden

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Attuel, MD, Principal Investigator — CNOM
Locations (37):
- France (37):
  - CHG, Abbeville
  - Hopital Privé, Antony
  - CH, Auxerre
  - CH, Avignon
  - Clinique de Bordeaux Cauderan, Bordeaux
  - CHU, Caen
  - CH, Castres
  - HIA Percy, Clamart
  - CH, Colmar
  - CH René Pleven, Dinan
  - CH, Dole
  - CH, Dunkirk
  - CH, Évreux
  - CH, Grenoble
  - CMC Parly II, Le Chesnay
  - CH, Le Havre
  - CH, Limoges
  - CH Saint Philibert, Lomme
  - Clinique de la Casamance, Marseille
  - Clinique Bouchard, Marseille
  - CHU La Timone, Marseille
  - CH, Martigues
  - CH, Metz
  - CHU, Montpellier
  - CH, Mulhouse
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Hopital Cardiologique du Haut Leveque, Pessac
  - Hopital Privé Claude Galien, Quincy-sous-Sénart
  - Polyclinique Saint Laurent, Rennes
  - CHU, Rennes
  - CHU, Rouen
  - CHU, Saint-Etienne
  - Institut Arnalt Tzanck, Saint-Laurent-du-Var
  - CMCO, Schiltigheim
  - CH, Thionville
  - CH Toulon, Toulon
  - CH, Valenciennes

REFERENCES:
- [Background] Fauchier L, Briand F, Soto FX, Quennelle F, Levy J, Darmon JP, Lellouche D, Lavergne T, Poret P, Pelade C, Babuty D. Management of atrial tachyarrhythmias: benefits of pacemaker diagnostics. Pacing Clin Electrophysiol. 2003 Jan;26(1P2):233-8. doi: 10.1046/j.1460-9592.2003.00023.x. PMID 12687819
- [Background] Camm AJ on behalf of the AFTherapy Study Group. The Atrial Fibrillation Therapy Study. Présentation orale au cours du Congrès de l'ESC à Stockholm, Septembre 2001.
- [Background] Fuster V, Ryden LE, Asinger RW, Cannom DS, Crijns HJ, Frye RL, Halperin JL, Kay GN, Klein WW, Levy S, McNamara RL, Prystowsky EN, Wann LS, Wyse DG; American College of Cardiology; American Heart Association; European Society of Cardiology; North American Society of Pacing and Electrophysiology. ACC/AHA/ESC guidelines for the management of patients with atrial fibrillation. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines and Policy Conferences (Committee to develop guidelines for the management of patients with atrial fibrillation) developed in collaboration with the North American Society of Pacing and Electrophysiology. Eur Heart J. 2001 Oct;22(20):1852-923. doi: 10.1053/euhj.2001.2983. No abstract available. PMID 11601835
- [Background] Tse HF, Lau CP, Ayers GM. Incidence and modes of onset of early reinitiation of atrial fibrillation after successful internal cardioversion, and its prevention by intravenous sotalol. Heart. 1999 Sep;82(3):319-24. doi: 10.1136/hrt.82.3.319. PMID 10455082
- [Background] Falk RH. Management of atrial fibrillation--radical reform or modest modification? N Engl J Med. 2002 Dec 5;347(23):1883-4. doi: 10.1056/NEJMe020137. No abstract available. PMID 12466514
- [Background] Van Gelder IC, Hagens VE, Bosker HA, Kingma JH, Kamp O, Kingma T, Said SA, Darmanata JI, Timmermans AJ, Tijssen JG, Crijns HJ; Rate Control versus Electrical Cardioversion for Persistent Atrial Fibrillation Study Group. A comparison of rate control and rhythm control in patients with recurrent persistent atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1834-40. doi: 10.1056/NEJMoa021375. PMID 12466507
- [Background] Wyse DG, Waldo AL, DiMarco JP, Domanski MJ, Rosenberg Y, Schron EB, Kellen JC, Greene HL, Mickel MC, Dalquist JE, Corley SD; Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM) Investigators. A comparison of rate control and rhythm control in patients with atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1825-33. doi: 10.1056/NEJMoa021328. PMID 12466506
- [Background] Hohnloser SH, Kuck KH, Lilienthal J. Rhythm or rate control in atrial fibrillation--Pharmacological Intervention in Atrial Fibrillation (PIAF): a randomised trial. Lancet. 2000 Nov 25;356(9244):1789-94. doi: 10.1016/s0140-6736(00)03230-x. PMID 11117910
- [Background] Hohnloser SH, Kuck KH. Randomized trial of rhythm or rate control in atrial fibrillation: the Pharmacological Intervention in Atrial Fibrillation Trial (PIAF). Eur Heart J. 2001 May;22(10):801-2. doi: 10.1053/euhj.2001.2596. No abstract available. PMID 11350085
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Defaye P, Dournaux F, Mouton E. Prevalence of supraventricular arrhythmias from the automated analysis of data stored in the DDD pacemakers of 617 patients: the AIDA study. The AIDA Multicenter Study Group. Automatic Interpretation for Diagnosis Assistance. Pacing Clin Electrophysiol. 1998 Jan;21(1 Pt 2):250-5. doi: 10.1111/j.1540-8159.1998.tb01098.x. PMID 9474682
- [Background] Andersen HR, Nielsen JC, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Long-term follow-up of patients from a randomised trial of atrial versus ventricular pacing for sick-sinus syndrome. Lancet. 1997 Oct 25;350(9086):1210-6. doi: 10.1016/S0140-6736(97)03425-9. PMID 9652562
- [Background] Connolly SJ, Kerr CR, Gent M, Roberts RS, Yusuf S, Gillis AM, Sami MH, Talajic M, Tang AS, Klein GJ, Lau C, Newman DM. Effects of physiologic pacing versus ventricular pacing on the risk of stroke and death due to cardiovascular causes. Canadian Trial of Physiologic Pacing Investigators. N Engl J Med. 2000 May 11;342(19):1385-91. doi: 10.1056/NEJM200005113421902. PMID 10805823
- [Background] Gillis AM, Connolly SJ, Lacombe P, Philippon F, Dubuc M, Kerr CR, Yee R, Rose MS, Newman D, Kavanagh KM, Gardner MJ, Kus T, Wyse DG. Randomized crossover comparison of DDDR versus VDD pacing after atrioventricular junction ablation for prevention of atrial fibrillation. The atrial pacing peri-ablation for paroxysmal atrial fibrillation (PA (3)) study investigators. Circulation. 2000 Aug 15;102(7):736-41. doi: 10.1161/01.cir.102.7.736. PMID 10942740
- [Background] Edvardson N. Efficacy of preventive pacing therapies in Paroxysmal Atrial Fibrillation - IV International meeting - Atrial Fibrillation 2001 : 161-164.
- [Background] Hoffmann E, Janko S, Steinbeck G and al. Onset scenarios of paroxysmal atrial fibrillation using new diagnostic pacemaker functions. Pacing Clin Electrophysiol. 2000 ; 23(4) : 656 (abstract).
- [Background] Hoffmann E, Janko S, Steinbeck G and al. Analysis of Onset Mechanisms of Paroxysmal Atrial Fibrillation through a Pacemaker with Continuous Monitoring Capabilities. Pacing Clin Electrophysiol. 2000 ; 23(4) : 656 (poster).
- [Background] Capucci A, Gropppi F, Ruiter J on behalf of the AFTherapy Study Group. Re-initiation of atrial Fibrillation Investigated Through pacemaker Focussed Diagnostics. Europace 2000 - Supplement 1.
- [Background] Tse HF, Lau CP, Ayers GM. Atrial pacing for suppression of early reinitiation of atrial fibrillation after successful internal cardioversion. Eur Heart J. 2000 Jul;21(14):1167-76. doi: 10.1053/euhj.1999.1991. PMID 10924300
- [Background] Lee JK, Yee R, Braney M, Stoop G, Begemann M, Dunne C, Klein GJ, Krahn AD, Van Hemel NM. Acute testing of the rate-smoothed pacing algorithm for ventricular rate stabilization. Pacing Clin Electrophysiol. 1999 Apr;22(4 Pt 1):554-61. doi: 10.1111/j.1540-8159.1999.tb00496.x. PMID 10234708
- [Background] Lau CP, Jiang ZY, Tang MO. Efficacy of ventricular rate stabilization by right ventricular pacing during atrial fibrillation. Pacing Clin Electrophysiol. 1998 Mar;21(3):542-8. doi: 10.1111/j.1540-8159.1998.tb00096.x. PMID 9558685
- [Background] Daoud EG, Weiss R, Bahu M, Knight BP, Bogun F, Goyal R, Harvey M, Strickberger SA, Man KC, Morady F. Effect of an irregular ventricular rhythm on cardiac output. Am J Cardiol. 1996 Dec 15;78(12):1433-6. doi: 10.1016/s0002-9149(97)89297-1. PMID 8970422
- [Background] Yee R, Meijer A and Winkler WB and al. Effect of Chronic Ventricular Rate Stabilization on Rate Irregularity in Patients with Permanent Atrial Fibrillation. Progress in Clinical Pacing - Rome 2002 : 52 (abstract)
- [Background] Pfaiffer L, Canby P, Navone A and al. Impact of Atrial Rhythm Diagnostics on Clinical Management. Europace Supplements 2002 ; 3 : A 152 (abstract).
- [Background] Gregoratos G, Abrams J, Epstein AE, Freedman RA, Hayes DL, Hlatky MA, Kerber RE, Naccarelli GV, Schoenfeld MH, Silka MJ, Winters SL. ACC/AHA/NASPE 2002 Guideline Update for Implantation of Cardiac Pacemakers and Antiarrhythmia Devices--summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/NASPE Committee to Update the 1998 Pacemaker Guidelines). J Am Coll Cardiol. 2002 Nov 6;40(9):1703-19. doi: 10.1016/s0735-1097(02)02528-7. No abstract available. PMID 12427427
- [Background] Jenkins LS, Bubien RS. Quality of life in patients with atrial fibrillation. Cardiol Clin. 1996 Nov;14(4):597-606. doi: 10.1016/s0733-8651(05)70307-6. PMID 8950060
- [Background] Carlioz R, Perrier E, Thomas O and al. Accuracy of atrial Tachyarrhythmia Monitoring in the Selection Device : Correlation with an External Holter Recording. Europace Suppl 2001 ; 2 : B199.
- [Background] Jenkins LS. Quality of life in Patients with Atrial Fibrillation. Circulation 1995 ; 92 (I) : 490 (abstract).
- [Background] Bubien RS, Knotts-Dolson SM, Plumb VJ, Kay GN. Effect of radiofrequency catheter ablation on health-related quality of life and activities of daily living in patients with recurrent arrhythmias. Circulation. 1996 Oct 1;94(7):1585-91. doi: 10.1161/01.cir.94.7.1585. PMID 8840848